CLINICAL TRIAL: NCT01860495
Title: Gingival Crevicular Fluid Bone Morphogenetic Protein - 2 Release Profile Following the Use of Modified Perforated Membrane Barriers in Localized Intrabony Defects (An in Vivo Study)
Brief Title: Gingival Crevicular Fluid Bone Morphogenetic Protein - 2 Release Profile Following the Use of Perforated Membrane
Acronym: MPM
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Y Gamal, professor of periodontology, Al-Azhar University
Other Study IDs: ahmedgamal
Record Dates: First submitted 2013-05-19; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Periodontal Pocket
Keywords: growth factors; periodontal pockets
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- perforated membrane group: perforated membrane group (G1- 15 sites)
  Interventions: Procedure: perforated membrane
- occlusive membrane group: occlusive collagen membrane that are tradetionally used in guided tissue regeneration , control occlusive group (G2-15 sites)
  Interventions: Procedure: G2

INTERVENTIONS:
Procedure: perforated membrane — perforated membrane that could give a chance for posetive contributionn of periosteal and gingival mesenchymal stem cells in periodontal regeneration
  Other Names: collagen membranes
  Groups: perforated membrane group
Procedure: G2 — tradetional occlusive collagen membrane
  Other Names: guided tissue membranes
  Groups: occlusive membrane group

SUMMARY:
One of the most important elements suggested to be provided through membrane perforations to augment regeneration are cell released growth factors from the overlying periosteal and gingival cells. A direct correlation could exist between the number of such cells and their available released growth factors. To test this assumption, this study was designed to evaluate levels of bone morphogenetic protein-2 in gingival crevicular fluid (GCF) during the early stages of healing for sites treated by MPM compared to that of the occlusive barrier membranes.

DETAILED DESCRIPTION:
The subjects were recruited consecutively from the list of patients seeking care for periodontal problems at the Department of Periodontology of the Faculty of Dental Medicine, Al Azhar University, Cairo, Egypt, between March 2012 to December 2012. The criteria implemented for patient inclusion were: 1) no systemic diseases which could influence the outcome of the therapy; 2) good compliance with the plaque control instructions following initial therapy; 3) teeth involved were all vital with score 0 mobility ; 4) each subject contributed matched pairs of two or three walled intrabony interproximal defects in premolar or molar teeth 5) the selected 2- or 3-wall intrabony defect depth ranged from 3-5 mm as detected in diagnostic periapical radiographs; 6) selected pocket depth (PD) ≥ 6 mm and clinical attachment level (CAL) ≥ 5 mm at the site of endosseous defect four weeks following initial cause-related therapy 7) endosseous radiographic defect angle ≤55 and ≥15 8) availability for the follow-up and maintenance program; 9) absence of periodontal treatment for the previous year; 10) absence of systemic medication or antibiotic treatment for the previous 6 months; 11) absence of a smoking habit and 12) absence of occlusal interferences. Pregnant females were excluded from participating in the study. Patients were also excluded from the study if they presented with opened interproximal contact, or inadequate compliance with the oral hygiene maintenance schedule. The experimental protocol was approved by the Ethical Committee of El Azhar University (OMD - 45 - 2012, clinical trial registration number: Al Azhar University 22-31). Research procedures were explained to all patients and they agreed to participate in the study and signed the appropriate informed consent form of Al Azhar University.

ELIGIBILITY:
Inclusion Criteria:

1. no systemic diseases which could influence the outcome of the therapy;
2. good compliance with the plaque control instructions following initial therapy;
3. teeth involved were all vital with score 0 mobility ;
4. each subject contributed matched pairs of two or three walled intrabony interproximal defects in premolar or molar teeth
5. the selected 2- or 3-wall intrabony defect depth ranged from 3-5 mm as detected in diagnostic periapical radiographs;
6. selected pocket depth (PD) ≥ 6 mm and clinical attachment level (CAL) ≥ 5 mm at the site of endosseous defect four weeks following initial cause-related therapy
7. endosseous radiographic defect angle ≤55 and ≥15
8. availability for the follow-up and maintenance program;
9. absence of periodontal treatment for the previous year;
10. absence of systemic medication or antibiotic treatment for the previous 6 months;
11. absence of a smoking habit and
12. absence of occlusal interferences.

Exclusion Criteria:

* Pregnant females were excluded from participating in the study.
* Patients were also excluded from the study if they presented with opened interproximal contact, or inadequate compliance with the oral hygiene maintenance schedule.

Ages: 31 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifteen non-smoking patients (8 males and 7 females) who were 31 to 51 years of age at the time of baseline examination (mean age 33.8 ± 6.1) with severe chronic periodontitis (Armitage 1999) participated in this prospective, randomized and blinded clinical trial. The subjects were recruited consecutively from the list of patients seeking care for periodontal problems at the Department of Periodontology of the Faculty of Dental Medicine, Al Azhar University, Cairo, Egypt, between March 2012 to December 2012. The experimental protocol was approved by the Ethical Committee of El Azhar University (OMD - 45 - 2012). Research procedures were explained to all patients and they agreed to participate in the study and signed the appropriate informed consent form of Al Azhar University.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
gingival cervicular fluid BMP-2 level | 30 days
  Using capillary tube (5 µl), gingival cervicular fluid (GCF) samples were collected (Sueda et al, 1969) by a single examiner (MA) who was masked to the attribution of the sites to MPM or OM. Following the isolation and drying of the selected site with cotton rolls, a fisher brand disposable micropipettes €, placed intrasulculary at the mesiofacial line angle of the selected site to a maximum depth of 2 mm below the gingival margin. Micropipettes were left in place until 5ul of fluid was collected. Gingival cervicular fluid (GCF) samples were collected one day, 3, 7, 14, 21, and 30 days after therapy and diluted in saline solution (50 µl) for bone morphogenetic protein-2 level evaluation. Samples were labeled, carried in a dark container and kept at -80 C until used.

SECONDARY OUTCOMES:
intrabony components (defect bony filling) | 9 months
  Clinical and radiographic measurements (pocket depth, attachement level, gingival index , plaque index, intrabony level) were reassessed at 3, 6, and 9 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, PhD, Principal Investigator — Al Azhar universty, faculty of dentistry, cairo, egypt; Mohamed M Aziz, BCH, Study Director — al azhar universty, cairo, egypt; Mohamed M Helmy, MSD, Study Director — al azhar universty; Vencint J Iacono, PhD, Study Chair — Stony Brook Uiversty
Locations (1):
- Al azhar universty, Cairo Governorate, Egypt, Egypt

REFERENCES:
- [Result] Gamal AY, Iacono VJ. Enhancing guided tissue regeneration of periodontal defects by using a novel perforated barrier membrane. J Periodontol. 2013 Jul;84(7):905-13. doi: 10.1902/jop.2012.120301. Epub 2012 Sep 24. PMID 23003916